CLINICAL TRIAL: NCT04059562
Title: Efficacy and Safety of Trifluridine/Tipiracil in Combination With Irinotecan as a Second Line Therapy in Patients With Cholangiocarcinoma
Brief Title: Trifluridine/Tipiracil in Combination With Irinotecan as a Second Line Therapy in Patients With Cholangiocarcinoma
Acronym: TRITICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-157
Record Dates: First submitted 2018-09-04; First posted 2019-08-16 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: Combination of Lonsurf® and Irinotecan in 28 patients with cholangiocarcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Combination of Lonsurf® and Irinotecan
  Interventions: Combination Product: Combination of Lonsurf® and Irinotecan

INTERVENTIONS:
Combination Product: Combination of Lonsurf® and Irinotecan — Trifluridine/Tipiracil (Lonsurf®) and Irinotecan
  * Trifluridine/Tipiracil will be administered at a dose of 25 mg/m2 / dose twice daily on days 1-5 followed by a 9-days recovery period from day 6 trough day 14 of each 14-days treatment cycle.
  * Irinotecan will be administered at the same time as Trifluridine/Tipiracil (Lonsurf®) on day 1 of each cycle at a dose of 180 mg/m2 / dose.

SUMMARY:
This is a prospective, single arm, open label, non-randomized, exploratory, multi-centre pilot study with median progression free survival as primary outcome.

In total 28 patients (including 3 calculated drop outs and invalid cases) with advanced cholangiocellular carcinoma after failure of a gemcitabine based first-line therapy will be enrolled at 5 centres.

To examine the efficacy of a combination therapy of Trifluridine/Tipiracil and Irinotecan in patients with advanced, non resectable or metastatic cholangio- and gallbladder carcinoma after failure to respond to a previous gemcitabine treatment.

The study will be accompanied by a translational research program:

Before treatment and after each radiological tumor assessment (Q6W) blood and stool will be collected and extensive panels of biomarkers will be accessed.

DETAILED DESCRIPTION:
This is a prospective, single arm, open label, non-randomized, exploratory, multi-centre pilot study with median progression free survival as primary outcome.

In total 28 patients (including 3 calculated drop outs and invalid cases) with advanced cholangiocellular carcinoma after failure of a gemcitabine based first-line therapy will be enrolled at 5 centres.

To examine the efficacy of a combination therapy of Trifluridine/Tipiracil and Irinotecan in patients with advanced, non resectable or metastatic cholangio- and gallbladder carcinoma after failure to respond to a previous gemcitabine treatment.

The study will be accompanied by a translational research program:

Before treatment and after each radiological tumor assessment (Q6W) blood and stool will be collected and extensive panels of biomarkers will be accessed.

Patients will be treated until radiological progression. In average this will be about 4 months. A follow up is planned every 3 months up to 6 months to asses life quality and progression data.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent incl. participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Histologically or cytologically confirmed, non-resectable, locally advanced or metastatic cholangiocarcinoma or gall bladder carcinoma
4. Measurable or assessable disease according to RECIST 1.1
5. Documented disease progression after prior gemcitabine or gemcitabine containing therapy. Examples of permitted therapies include, but are not limited to: a) Single agent gemcitabine); b) Any gemcitabine-based regimen, with or without maintenance gemcitabine
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Ability to take medications orally
8. Adequate blood count, liver-enzymes, and renal function:

   * Absolute neutrophil count (ANC) > 1,500 cells/μL without the use of hematopoietic growth factors; and Platelet count ≥ 100 x 109/L (>100,000 per mm3) and Hemoglobin > 9 g/dL (blood transfusions are permitted for patients with hemoglobin levels below 9 g/dL)
   * Serum total bilirubin ≤ 1.5x upper normal limit (ULN) (biliary drainage is allowed for biliary obstruction; elevated bilirubin should be caused by obstruction not impaired liver function as assessed by albumin and international normalised ratio (INR) values):
   * Albumin levels ≥ 3.0 g/dL
   * Patients not receiving therapeutic anticoagulation must have an INR< 1.5 ULN and partial thromboplastin time (PTT) < 1.5 ULN within 7 days prior to inclusion. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of inclusion.
   * aspartate aminotransferase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) ≤ 5 x institutional upper limit of normal
   * Serum Creatinine ≤ 1.5 x ULN and a calculated glomerular filtration rate ≥ 30 mL per minute Adequate renal and bone marrow function
9. In case of liver cirrhosis: Child-Pugh A
10. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control

Exclusion Criteria:

1. Age < 18 years
2. Central nerve system (CNS) metastases
3. Active, uncontrolled infection
4. Additional malignancy within the past 2 years (except adequately treated in-situ carcinoma of the cervix or non-melanoma skin cancer)
5. Clinically significant gastrointestinal disorders including bleeding, inflammation, occlusion, or diarrhea > grade 1
6. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
7. Known hypersensitivity to Trifluridine/Tipiracil or Camptothecin (CPT)-11 or their components
8. Medication that is known to interfere with any of the agents applied in the trial
9. Pregnancy or lactating female
10. Prior partial or total gastrectomy
11. Previous radio- or radiochemotherapy, previous transarterial chemoembolisation (TACE), radiofrequency ablation (RFA) or selective intraarterial radiotherapy (SIRT) within 3 months prior to inclusion (except radiation for bone metastases)
12. Patients who might be dependent on the sponsor, site or the investigator
13. Patients who have been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
14. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a German drug law (AMG)].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Median progression free survival (PFS) | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Median progression free survival (PFS)

SECONDARY OUTCOMES:
Progression-free survival rate | At 4 months
  Progression-free survival rate @ 4 months defined as the proportion of patients with non-progressive disease 4 months after inclusion by intention to treat analysis
Median overall survival | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Median overall survival
Response according to RECIST 1.1 | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Proportion of patients with an objective response according to RECIST 1.1
Safety (type, grade and frequency of Adverse Events (AEs)/Serious Adverse Events (SAEs)) | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Safety (type, grade and frequency of AEs/SAEs)
Quality of life - European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-30) | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Analysis of quality of life (EORTC QLQ-30)
Quality of life - EuroQol-5Dimensions-3Levels (EQ-5D-5L) questionnaires | through study completion, an average of 1 year (~4 months intervention + 6 months Follow Up)
  Analysis of quality of life (EQ-5D-5L questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Roderburg, Prof., Principal Investigator — Klinik für Gastroenterologie, Hepatologie und Infektiologie Universitätsklinikum Düsseldorf
Locations (1):
- Klinik für Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plentz RR, Malek NP. Clinical presentation, risk factors and staging systems of cholangiocarcinoma. Best Pract Res Clin Gastroenterol. 2015 Apr;29(2):245-52. doi: 10.1016/j.bpg.2015.02.001. Epub 2015 Feb 14. PMID 25966425
- [Background] Muller RK. [Documentation of forensic-chemical studies on punched cards]. Dtsch Z Gesamte Gerichtl Med. 1966;58(1):65-75. No abstract available. German. PMID 5966423
- [Background] Blechacz BR, Gores GJ. Cholangiocarcinoma. Clin Liver Dis. 2008 Feb;12(1):131-50, ix. doi: 10.1016/j.cld.2007.11.003. PMID 18242501
- [Background] Okusaka T, Nakachi K, Fukutomi A, Mizuno N, Ohkawa S, Funakoshi A, Nagino M, Kondo S, Nagaoka S, Funai J, Koshiji M, Nambu Y, Furuse J, Miyazaki M, Nimura Y. Gemcitabine alone or in combination with cisplatin in patients with biliary tract cancer: a comparative multicentre study in Japan. Br J Cancer. 2010 Aug 10;103(4):469-74. doi: 10.1038/sj.bjc.6605779. Epub 2010 Jul 13. PMID 20628385
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Walter T, Horgan AM, McNamara M, McKeever L, Min T, Hedley D, Serra S, Krzyzanowska MK, Chen E, Mackay H, Feld R, Moore M, Knox JJ. Feasibility and benefits of second-line chemotherapy in advanced biliary tract cancer: a large retrospective study. Eur J Cancer. 2013 Jan;49(2):329-35. doi: 10.1016/j.ejca.2012.08.003. Epub 2012 Sep 1. PMID 22947649
- [Background] Lamarca A, Hubner RA, David Ryder W, Valle JW. Second-line chemotherapy in advanced biliary cancer: a systematic review. Ann Oncol. 2014 Dec;25(12):2328-2338. doi: 10.1093/annonc/mdu162. Epub 2014 Apr 25. PMID 24769639
- [Background] Guion-Dusserre JF, Lorgis V, Vincent J, Bengrine L, Ghiringhelli F. FOLFIRI plus bevacizumab as a second-line therapy for metastatic intrahepatic cholangiocarcinoma. World J Gastroenterol. 2015 Feb 21;21(7):2096-101. doi: 10.3748/wjg.v21.i7.2096. PMID 25717243
- [Background] Petrelli F, Inno A, Ghidini A, Rimassa L, Tomasello G, Labianca R, Barni S; GISCAD (Gruppo Italiano per lo Studio dei Carcinomi dell'Apparato Digerente) and Cremona Hospital. Second line with oxaliplatin- or irinotecan-based chemotherapy for gemcitabine-pretreated pancreatic cancer: A systematic review. Eur J Cancer. 2017 Aug;81:174-182. doi: 10.1016/j.ejca.2017.05.025. PMID 28633088
- [Background] Vanhoefer U, Harstrick A, Achterrath W, Cao S, Seeber S, Rustum YM. Irinotecan in the treatment of colorectal cancer: clinical overview. J Clin Oncol. 2001 Mar 1;19(5):1501-18. doi: 10.1200/JCO.2001.19.5.1501. PMID 11230497
- [Background] Burris HA 3rd, Fields SM. Topoisomerase I inhibitors. An overview of the camptothecin analogs. Hematol Oncol Clin North Am. 1994 Apr;8(2):333-55. PMID 8040144
- [Background] Toffoli G, Cecchin E, Corona G, Boiocchi M. Pharmacogenetics of irinotecan. Curr Med Chem Anticancer Agents. 2003 May;3(3):225-37. doi: 10.2174/1568011033482477. PMID 12769780
- [Background] Irinotecan. 2025 Jan 15. Drugs and Lactation Database (LactMed(R)) [Internet]. Bethesda (MD): National Institute of Child Health and Human Development; 2006-. Available from http://www.ncbi.nlm.nih.gov/books/NBK500877/ PMID 29999936
- [Background] Emura T, Murakami Y, Nakagawa F, Fukushima M, Kitazato K. A novel antimetabolite, TAS-102 retains its effect on FU-related resistant cancer cells. Int J Mol Med. 2004 Apr;13(4):545-9. PMID 15010854
- [Background] Emura T, Suzuki N, Yamaguchi M, Ohshimo H, Fukushima M. A novel combination antimetabolite, TAS-102, exhibits antitumor activity in FU-resistant human cancer cells through a mechanism involving FTD incorporation in DNA. Int J Oncol. 2004 Sep;25(3):571-8. PMID 15289858
- [Background] Farshidfar F, Zheng S, Gingras MC, Newton Y, Shih J, Robertson AG, Hinoue T, Hoadley KA, Gibb EA, Roszik J, Covington KR, Wu CC, Shinbrot E, Stransky N, Hegde A, Yang JD, Reznik E, Sadeghi S, Pedamallu CS, Ojesina AI, Hess JM, Auman JT, Rhie SK, Bowlby R, Borad MJ; Cancer Genome Atlas Network; Zhu AX, Stuart JM, Sander C, Akbani R, Cherniack AD, Deshpande V, Mounajjed T, Foo WC, Torbenson MS, Kleiner DE, Laird PW, Wheeler DA, McRee AJ, Bathe OF, Andersen JB, Bardeesy N, Roberts LR, Kwong LN. Integrative Genomic Analysis of Cholangiocarcinoma Identifies Distinct IDH-Mutant Molecular Profiles. Cell Rep. 2017 Jun 27;19(13):2878-2880. doi: 10.1016/j.celrep.2017.06.008. PMID 28658632
- [Background] Roderburg C, Urban GW, Bettermann K, Vucur M, Zimmermann H, Schmidt S, Janssen J, Koppe C, Knolle P, Castoldi M, Tacke F, Trautwein C, Luedde T. Micro-RNA profiling reveals a role for miR-29 in human and murine liver fibrosis. Hepatology. 2011 Jan;53(1):209-18. doi: 10.1002/hep.23922. Epub 2010 Oct 1. PMID 20890893
- [Background] Lin XJ, Chong Y, Guo ZW, Xie C, Yang XJ, Zhang Q, Li SP, Xiong Y, Yuan Y, Min J, Jia WH, Jie Y, Chen MS, Chen MX, Fang JH, Zeng C, Zhang Y, Guo RP, Wu Y, Lin G, Zheng L, Zhuang SM. A serum microRNA classifier for early detection of hepatocellular carcinoma: a multicentre, retrospective, longitudinal biomarker identification study with a nested case-control study. Lancet Oncol. 2015 Jul;16(7):804-15. doi: 10.1016/S1470-2045(15)00048-0. Epub 2015 Jun 15. PMID 26088272
- [Background] Cao J, Sun L, Li J, Zhou C, Cheng L, Chen K, Yan B, Qian W, Ma Q, Duan W. A novel three-miRNA signature predicts survival in cholangiocarcinoma based on RNA-Seq data. Oncol Rep. 2018 Sep;40(3):1422-1434. doi: 10.3892/or.2018.6534. Epub 2018 Jun 27. PMID 29956786
- [Background] Meirow Y, Baniyash M. Immune biomarkers for chronic inflammation related complications in non-cancerous and cancerous diseases. Cancer Immunol Immunother. 2017 Aug;66(8):1089-1101. doi: 10.1007/s00262-017-2035-6. Epub 2017 Jul 3. PMID 28674756
- [Background] Yu LX, Schwabe RF. The gut microbiome and liver cancer: mechanisms and clinical translation. Nat Rev Gastroenterol Hepatol. 2017 Sep;14(9):527-539. doi: 10.1038/nrgastro.2017.72. Epub 2017 Jul 5. PMID 28676707
- [Background] Schwarz R, Hinz A. Reference data for the quality of life questionnaire EORTC QLQ-C30 in the general German population. Eur J Cancer. 2001 Jul;37(11):1345-51. doi: 10.1016/s0959-8049(00)00447-0. PMID 11435063
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] King MT. The interpretation of scores from the EORTC quality of life questionnaire QLQ-C30. Qual Life Res. 1996 Dec;5(6):555-67. doi: 10.1007/BF00439229. PMID 8993101
- [Background] Hjermstad MJ, Fayers PM, Bjordal K, Kaasa S. Using reference data on quality of life--the importance of adjusting for age and gender, exemplified by the EORTC QLQ-C30 (+3). Eur J Cancer. 1998 Aug;34(9):1381-9. doi: 10.1016/s0959-8049(98)00136-1. PMID 9849421
- [Background] Uwer L, Rotonda C, Guillemin F, Miny J, Kaminsky MC, Mercier M, Tournier-Rangeard L, Leonard I, Montcuquet P, Rauch P, Conroy T. Responsiveness of EORTC QLQ-C30, QLQ-CR38 and FACT-C quality of life questionnaires in patients with colorectal cancer. Health Qual Life Outcomes. 2011 Aug 22;9:70. doi: 10.1186/1477-7525-9-70. PMID 21859485
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Pickard AS, Wilke CT, Lin HW, Lloyd A. Health utilities using the EQ-5D in studies of cancer. Pharmacoeconomics. 2007;25(5):365-84. doi: 10.2165/00019053-200725050-00002. PMID 17488136
- [Derived] Kehmann L, Berres ML, Gonzalez-Carmona M, Modest DP, Mohr R, Wree A, Venerito M, Strassburg C, Keitel V, Trautwein C, Luedde T, Roderburg C. Study protocol of an open-label, single arm phase II trial investigating the efficacy and safety of Trifluridine/Tipiracil combined with irinotecan as a second line therapy in patients with cholangiocarcinoma (TRITICC). BMC Cancer. 2023 May 22;23(1):470. doi: 10.1186/s12885-023-10972-6. PMID 37217885